CLINICAL TRIAL: NCT04129567
Title: Transnasal Therapy for Acute Migraine Attack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00166706
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Migraine Disorders
Keywords: Trans-nasal; acute; migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Humidified oxygen (Experimental): Delivering humidified oxygen at 15 liters per minute through the nose and noting the change in primary and secondary outcome variables at 2 hours and 24 hours.
  Interventions: Other: Humidified oxygen
- Dry air (Experimental): Delivering dry air at 15 liters per minute through the nose and noting the change in primary and secondary outcome variables at 2 hours and 24 hours.
  Interventions: Other: Dry air
- Humidified air (Placebo Comparator): Delivering humidified air at 15 liters per minute through the nose and noting the change in primary and secondary outcome variables at 2 hours and 24 hours.
  Interventions: Other: Humidified air
- Dry oxygen (Active Comparator): Delivering dry oxygen at 15 liters per minute through the nose and noting the change in primary and secondary outcome variables at 2 hours and 24 hours.
  Interventions: Other: Dry oxygen

INTERVENTIONS:
Other: Humidified oxygen — Delivering humidified oxygen at 15 liters per minute through the nose in a blinded fashion using a nasal cannula.
  Arms: Humidified oxygen
Other: Dry oxygen — Delivering dry oxygen at 15 liters per minute through the nose in a blinded fashion using a nasal cannula.
  Arms: Dry oxygen
Other: Humidified air — Delivering humidified air at 15 liters per minute through the nose in a blinded fashion using a nasal cannula.
  Arms: Humidified air
Other: Dry air — Delivering dry air at 15 liters per minute through the nose in a blinded fashion using a nasal cannula.
  Arms: Dry air

SUMMARY:
Migraine is a significant health problem in the United States with 34 million Americans suffering from migraine attacks every year. High-flow oxygen has been successfully used in several clinical studies. Vasoconstriction of blood vessels in the scalp has been proposed as a possible mechanism of action. Some researchers have suggested that the cooling effect of high-flow dry oxygen may be in part responsible for the pain relief. The main objective is to test the hypothesis that the pain relief obtained during high-flow trans-nasal gas therapy is due to the cooling effect of dry gas on the nasal mucosa. The study entails recruiting patients from a headache clinic, being escorted to the Institute for Clinical and Translational Research (ICTR) Johns Hopkins Bayview and randomized into different groups (humidified oxygen, dry air, humidified air and dry oxygen). Eventually, patients will be asked to fill out a questionnaire on pain, nausea, sound and light sensitivity graded on a scale of 1-10. Readings are noted at baseline, 15 mins, 2 hours and 24 hours post-therapy.

DETAILED DESCRIPTION:
Migraine headaches are associated with significant impairment of quality of life and loss of productivity. High-flow oxygen has been successfully used in several clinical trials and vasoconstriction of blood vessels has been postulated as a possible mechanism. Some researchers have suggested that the cooling effect of high-flow dry oxygen may be in part responsible for the pain relief.The main objective is to test the hypothesis that the pain relief obtained during high-flow intra-nasal gas therapy is due to the cooling effect of dry gas on the nasal mucosa. Participants for this study are recruited from the pool of patients who are already scheduled to attend the headache clinic staffed by the principal investigator. The PI will recruit patients at the Headache Clinic. The patients are escorted to the Clinical Trials Unit (CTU) at the Johns Hopkins Bayview where therapy its provided and will be asked to fill out a questionnaire on pain, nausea, sound and light sensitivity using a visual analog score (VAS) for each symptom on a scale of 1-10. The patients will be randomized to either humidified oxygen, dry air, humidified air or dry oxygen. Patients will be asked to submit readings at the end of therapy, at 2 hours and 24 hours post-therapy. Treatment failure is defined as persistent headache despite treatment with oxygen or air. Participants will be removed from the trial if participants prematurely terminate therapy.

The investigators believe that using a total sample size of 45 patients, the investigators will be able to show a statistically significant difference of >2 point change in the VAS pain score reduction between the two treatment groups with a confidence of 80%. No risk were reported in prior studies involving >100 patients and >500 episodes of treatment with air or oxygen. Because of the (at least 2 and 1/2 hour) delay in initiating standard of care treatments, subjects may experience a longer duration and/or intensity of pain from the headache than regular standards of care i.e., sooner. Participants will be reimbursed for participation in this study which will compensate travel and parking.

ELIGIBILITY:
Inclusion Criteria:

* Migraine diagnosis of at least 1 year
* Migraine attacks between 1 and 15 per month
* Onset of first migraine < 50 years of age
* Migraine prophylaxis medication unchanged for 3 months prior to enrollment
* Meets international classification for headache disorders criteria for diagnosis of episodic migraine with or without aura
* Able to attend a short treatment session within half hour of onset of headache.

Exclusion Criteria:

* Known oxygen dependency to maintain arterial oxygen saturation (SaO2) >95%
* Known marked nasal septal deviation
* Recurrent epistaxis or chronic Rhino-Sinusitis
* Concurrent sinus/intranasal surgery
* Unable to fully understand the consent process and informed consent due to either language barriers or mental capacity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
change in pain score as assessed on the VAS scale | 2 hours and 24 hours
  Graded on a scale of 1-10 where higher scores mean more pain.

SECONDARY OUTCOMES:
change in nausea score as assessed on the VAS scale | 2 hours and 24 hours
  Graded on a scale of 1-10 where higher scores mean more nausea.
change in light sensitivity score as assessed on the VAS scale | 2 hours and 24 hours
  Graded on a scale of 1-10 where higher scores mean more light sensitivity.
change in sound sensitivity score as assessed on the VAS scale | 2 hours and 24 hours
  Graded on a scale of 1-10 where higher scores mean more sound sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Nauman Tariq, MD, Principal Investigator — Johns Hopkins Neurology (Bayview)
Locations (1):
- Clinical Trials Unit, Johns Hopkins Bayview (JHU ICTR), Baltimore, Maryland, United States

REFERENCES:
- [Derived] Shah R, Assis F, Narasimhan B, Khachadourian V, Zhou S, Tandri H, Tariq N. Trans-nasal high-flow dehumidified air in acute migraine headaches: A randomized controlled trial. Cephalalgia. 2021 Aug;41(9):968-978. doi: 10.1177/0333102421997766. Epub 2021 Feb 25. PMID 33631965